CLINICAL TRIAL: NCT03853577
Title: Characterization of Altered Waking States of Consciousness in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PSICON-132
Record Dates: First submitted 2019-01-10; First posted 2019-02-25 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2020-04

CONDITIONS: Altered Waking States of Consciousness in Healthy Humans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Active Comparator)
  Interventions: Other: TMS/EEG
- Placebo (Placebo Comparator)
  Interventions: Other: TMS/EEG

INTERVENTIONS:
Other: TMS/EEG — navigated TMS/high-density(hd)-EEG to directly stimulate defined cortical areas and investigate quantitatively the level of consciousness in psilocybin-induced altered brain states

SUMMARY:
Altered waking states of consciousness and its underlying functional organization have gained increasing interest in recent years, i.e. in identifying the neural basis of consciousness. To overcome fundamental shortcomings of current methods to objectively assess the level of consciousness, the investigators propose here to apply a novel and empirically validated measure called 'perturbational complexity index' (PCI) based on the integrated information theory (IIT). This involves a combination of transcranial magnetic stimulation (TMS) and highdensity electroencephalography (hd-EEG) to measure electrocortical responses as distributed cerebral interactions ('integration') and spatiotemporal pattern ('information'). Given the finding of subjectively expanded consciousness as induced here by psilocybin, the investigators hypothesize that the PCI may be higher in such states. This will be the first TMS/hd-EEG study to investigate quantitatively the level of consciousness in a pharmacologically altered waking state of consciousness.

DETAILED DESCRIPTION:
In this study the investigators will apply navigated TMS/high-density(hd)-EEG to directly stimulate defined cortical areas and investigate quantitatively the level of consciousness in psilocybin-induced altered brain states. For this purpose, PCI is the primary outcome in psilocybin versus placebo condition. Given the findings and the subjective feeling of an 'expanded' consciousness in such states, the investigators primarily hypothesize that psilocybin will induce a higher PCI as compared to placebo in TMS/hd-EEG measurements over all targeted cortical areas in the acute phase of treatment (80 minutes after substance intake). Measurements will be done over the premotor cortex (Brodmann-Areal BA06), the midline sensorimotor cortex (BA04) and the superior occipital gyrus/cuneus (BA19) and may be related to the experience of an altered sense of self, e.g. measures of selflessness and egodissolution.

This study further seeks to characterize the effects of psilocybin compared to placebo on resting state EEG. To this aim, the current source density and the lagged phase synchronization of neuronal oscillations across distributed brain regions will be computed and correlated to reproduce interesting results in a recent work of Kometer and colleagues. More specifically, psilocybin decreased the current source density of neuronal oscillations within a neural network comprising the anterior and posterior cingulate cortices and parahippocampal regions. Even more, psilocybin-induced insightfulness and spiritual experience correlated with the lagged phase synchronization of delta oscillations between the retrosplenial cortex, the parahippocampus and the lateral orbitofrontal area, showing evidence for a direct association of spatiotemporal neuronal mechanism with enhanced insight into life and existence. The investigators therefore hypothesize that current source density of neuronal oscillations within the cingulate cortices and the parahippocampal regions (1.5-20 Hz) will be decreased and the lagged-phase synchronization of delta oscillations (1.5-4 Hz) between the retrosplenial cortex, the parahippocampus and the lateral orbitofrontal area will be correlated to insightfulness.

Additionally, psychometric assessment of the sense of self, of perceptual alterations and of mood will be conducted before and after each TMS session (Hood's Mysticism-Scale; 5-Dimensional Altered States of Consciousness Rating Scale; Positive and Negative Affect Schedule). the investigators expect to find a relationship between substance induced changes in perception and mood as indexed by these questionnaires.

Furthermore, the investigators will be conducting a probabilistic learning task (emotLearn) to examine the computational processes behind the interaction between reward learning and subconscious versus conscious emotional processing to estimate how emotional stimuli affect the learning rate in psilocybin compared to placebo condition. The investigators hypothesize that psilocybin decreases the conscious and subconscious learning rate by attenuating the processing of emotional cues.

The study design will be randomized, double-blind, placebo-controlled with one-time application of a single dose for each substance (moderate psilocybin dose of 20mg versus mannitol), within-subject and single center at the Psychiatrische Universitätsklinik Zurich. The number of participants is 25 healthy subjects as determined by power analysis. Inclusion criteria are healthy male or female volunteers aged 18-40 years. Exclusion criteria are personal and family history of major psychiatric disease (e.g. major depression, bipolar disorder, psychotic disorder) as defined in the DSM-V, any major medical condition (e.g. neurologic, cardiovascular, metabolic disease), family history of seizure disorder, current psychopharmacological treatment or pregnant respectively breastfeeding women. The study comprises a total of 3 visits in 3 weeks - 1 screening visit and 2 investigational visits and a written follow-up 12 weeks after the last investigational visit per participant. On the investigational visits participants will receive placebo or psilocybin in a randomized and counterbalanced order. The screening visit consists of a psychiatric assessment, physical examination, routine lab/toxicology, electrocardiogram (ECG), EEG and cranial T1 weighted magnetic resonance tomography (MRT). Study duration will be 2-3 years.

The research project was approved by the local ethics committee (KEK Zurich) in December 2018 as "Other clinical trial" as specified in the "Ordinance on Clinical Trials in Human Research" (KlinV, Chapter 2) without health-related intervention or investigational Medical Product (IMP) [25], Category B.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers aged 18-40 years

Exclusion Criteria:

* Personal and family history of major psychiatric disease (e.g. major depression, bipolar disorder, psychotic disorder) as defined in the DSM-V
* Any major medical condition (e.g. neurologic, cardiovascular, metabolic disease), family history of seizure disorder
* Current psychopharmacological treatment / use of medication
* Pregnant or breastfeeding women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
Assessment of change of the 'perturbational complexity index' (PCI) in psilocybin compared to placebo condition in healthy humans as indexed by TMS/EEG respones | First investigational visit at week 1, second investigational visit at week 3
  Application of navigated TMS/EEG over the premotor cortex (Brodmann-Area BA06), the midline sensorimotor cortex (BA04) and the superior occipital gyrus/cuneus (BA19)

SECONDARY OUTCOMES:
Assessment of change of the learning rate in a probabilistic learning task in psilocybin compared to placebo condition | First investigational visit at week 1, second investigational visit at week 3
  Application of a probabilistic learning task to examine the computational processes behind the interaction between reward learning and subconscious/conscious emotional processing
Assessment of change of the effect of psilocybin compared to placebo condition on all frequency bands of resting state EEG | First investigational visit at week 1, second investigational visit at week 3
  Resting state EEG will be collected before and after TMS/EEG sessions. This data will be used to calculate the 'current source density' (CSD) and the 'laged phase synchronization', serving as biomarkers for insightfulness and spiritual experience. More specifically, eight frequency will be investigated: delta (1.5-4 Hz), theta (4-8 Hz), alpha1 (8-10.5 Hz), alpha2 (10.5-13 Hz), beta1 (13-20 Hz), beta2 (20-30 Hz), gamma1 (30-45 Hz), gamma2 (55- 100 Hz)
Psychometric assessment of change of the sense of self, of perceptual alterations and of mood in psilocybin compared to placebo condition (1) | First investigational visit at week 1, second investigational visit at week 3
  Application of the 'Hood's Mysticism-Scale' (MS) before and after TMS/EEG sessions. The revised and validated Hood's Mysticism-Scale describes a measure of reported mystical experience. Items on this scale are positively and negatively expressed, and they comprise two major factors, a general mystical experience factor and a religious interpretation factor. The scale ranges from +4 (very correct) to -4 (very wrong)
Psychometric assessment of change of the sense of self, of perceptual alterations and of mood in psilocybin compared to placebo condition (2) | First investigational visit at week 1, second investigational visit at week 3
  Application of the '5-Dimensional Altered States of Consciousness Rating Scale' (5D-ASC) before and after TMS/EEG sessions. It is a retrospectively assessed questionnaire to measure subjective experiences of altered states of consciousness. It contains 94 items which are formulated as a visual analog scale. It contains five primary dimensions a global dimension of altered states of onsciousness: Oceanic boundlessness (OSE), Dread of Ego dissolution (AIA), Visionary restructuralization (VUS), Auditive alteration (AVE) and Vigilance reduction (VIR). The first-mentioned three dimensions correlate with each other and form a global dimension (G-ABZ). The visual analog scale (VAS) ranges from 0 (not perceived) to 10 (very strongly perceived)
Psychometric assessment of change of the sense of self, of perceptual alterations and of mood in psilocybin compared to placebo condition (3) | First investigational visit at week 1, second investigational visit at week 3
  Application of the 'Positive and Negative Affect Schedule' (PANAS) before and after TMS/EEG sessions. This is a questionnaire with 20 items about positive and negative affect. They reflect dispositional dimensions. A high score on negative affect is coupled with subjective distress and unpleasurable engagement. Positive affect represents the extent to which an individual experiences pleasurable engagement with the environment. The scale ranges from +2 (very strong) to -2 (very weak)
Psychometric assessment of change of the sense of self, of perceptual alterations and of mood in psilocybin compared to placebo condition (4) | First investigational visit at week 1, second investigational visit at week 3
  Application of the the 'Interoception Rating Scale' (IRS) before and after TMS/EEG sessions. The Interoception Rating Scale is a measure of numerous facets of interoception (e.g. intensity of heartbeat or breathing) with 14 items. Dial ratings on the VAS can range from 0 (none) to 100 (most intense)

CONTACTS AND LOCATIONS:
Overall Officials: Franz X. Vollenweider, Prof, MD, Principal Investigator — Psychiatric Hospital, University of Zurich
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ip CT, Olbrich S, de Bardeci M, Monn A, Ort A, Smallridge JW, Vollenweider F. Psilocybin-induced alterations in EEG power, connectivity and network dynamics in healthy subjects: Correlations with subjective experience and implications for therapeutic applications. Prog Neuropsychopharmacol Biol Psychiatry. 2026 Jan 27:111626. doi: 10.1016/j.pnpbp.2026.111626. Online ahead of print. PMID 41611012